CLINICAL TRIAL: NCT04547192
Title: Improving Initial Management of the Injured at Ghanaian District and Regional Hospitals With a Trauma Intake Form
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kwame Nkrumah University of Science and Technology (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: R21TW011685 (NIH); 1R21TW011685-01 (NIH)
Record Dates: First submitted 2020-09-03; First posted 2020-09-14 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Behavior Problem
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized clinical trial with introduction of the TIF at 8 hospitals sequentially, with start times randomized by stepped-wedge design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre TIF introduction (No Intervention): Emergency Health Service prior to introduction of TIF.
- Post introduction of TIF (Experimental): Emergency Health Service after introduction of TIF.
  Interventions: Other: Improving initial care of the injured

INTERVENTIONS:
Other: Improving initial care of the injured — Improvement in Care Processes
  Arms: Post introduction of TIF

SUMMARY:
Brief Summary: Improving care of the injured (trauma care) is a way to the large burden of injury in low- and middle-income countries. The important initial period of trauma care is often chaotic and prone to errors. The World Health Organization created a Trauma Care Checklist (TCC), which improved key performance indicators of care at tertiary hospitals but encountered factors which decreased its uptake. The investigators propose the use of a model Trauma Intake Form (TIF) with potential to achieve the benefits of the TCC, but with automatic usage and with accompanying improvements in documentation for key elements of care. It is especially oriented for smaller hospitals. The investigators propose a pragmatic randomized clinical trial with introduction of the TIF at 8 hospitals sequentially, with start times randomized by stepped-wedge design. Specifically, the investigators aim to determine the effectiveness the TIF to function as a checklist for increasing the appropriate use of key performance indicators during care of the injured in emergency units of non-tertiary hospitals in Ghana, as assessed by independent observers; to determine the percent of injured patients with adequate data on initial assessment before vs. after introduction of the TIF in emergency units of non-tertiary hospitals in Ghana; and to increase the capacity of the Kwame Nkrumah University of Science and Technology and the network of non-tertiary hospitals in southern Ghana to undertake high-quality trauma care research, including clinical trials.

DETAILED DESCRIPTION:
Background: Injuries constitute an important public health problem in Ghana and other low- and middle-income countries (LMIC). The large burden of injury can be reduced by strengthening the process of care (1). The period of initial assessment and care of the injured has been identified as having the potential for significant errors (2, 3). Quality improvement efforts can reduce these errors (4, 5).

A systematic approach to the initial assessment and care of the injured ensures early detection of life-threatening conditions, prompting timely performance of necessary interventions (6, 7). The WHO Trauma Care Checklist (TCC), specifically developed for the early assessment and care of injured patients, led to improvements in key performance indicators of care as well as a decrease in mortality (1). Despite the usefulness of checklists in surgical practice, many countries report low usage rates (8-11). One unique barrier with the TCC is its application at the end of the initial trauma assessment, by which time some members of the trauma team may have left (12). Other approaches that would trigger more automatic use of the checklist might achieve the objectives of the TCC while improving compliance to its use. The Trauma Intake Form (TIF) to be tested in this study has been designed to achieve this goal.

An additional functionality of the TIF is improving data recording for both better immediate clinical care and better ability to conduct quality improvement programs. Data elements needed for this purpose were created through a Delphi process to develop a set of key performance indicators that were deemed to be accurate proxies of quality trauma care, simple to measure and feasible to collect at non-tertiary hospitals of LMICs (13). The TIF was created as a means of operationalizing key performance indicators by building them into the clinical chart of injured patients undergoing initial care in emergency units.

The extent to which a systematic approach is employed in the initial assessment of injured patients arriving at emergency units of district and regional hospitals in Ghana is unknown. With successful training of emergency health service providers in the use of the TIF and its subsequent adoption, improvements in systematic assessment and care of the injured in these hospitals can be achieved.

Specific aim 1. To determine the effectiveness of the TIF to function as a checklist for increasing the appropriate use of key performance indicators during care of the injured in emergency units in district and regional hospitals in Ghana, as assessed by independent observers.

Hypothesis: The TIF will increase the appropriate use of key performance indicators by significant and clinically meaningful levels. For example, we expect the TIF to increase the percent of all injured patients whose blood pressure is checked at arrival by a minimum of 8%, and increase the percent of those with heart rate checked by a minimum of 8%. For seriously injured patients, we expect the TIF to improve the achievement of additional key performance indicators by clinically meaningful levels. For example, we expect the TIF to increase the percent of patients with chest examination by a minimum of 8%, increase the percent of patients with hemoperitoneum ruled out by a minimum of 12%, and improve the percent of patients with examination of all distal pulses by a minimum of 13%.

Specific aim 2. To determine the percent of injured patients with adequate data on initial assessment before vs. after introduction of the TIF in emergency units in district and regional hospitals in Ghana.

Hypothesis. The TIF will increase documentation of important clinical data on injured patients (including all of the following: time of injury, mechanism of injury, respiratory rate at presentation, heart rate at presentation, blood pressure at presentation, consciousness level at presentation, temperature at presentation, and time of disposition) by at least 5%.

Specific aim 3. To increase the capacity of the Kwame Nkrumah University of Science and Technology and the network of district and regional hospitals in to undertake high-quality trauma care research, including clinical trials.

Methods A pragmatic randomized clinical trial will be carried out at 8 district and regional hospitals in Ghana. The intervention to be tested is the TIF to be used in recording information about injured patients during their initial assessment and care and which is designed to decrease omission of critical steps in care and so to improve care and also record keeping.

The unit of randomization will be hospitals and a stepped-wedge design will be used to select which hospitals will start use of the TIF at what time. We have select eight hospitals across four regions in Ghana to represent district or regional hospitals with more than adequate flow of injured patients (≥75 patients per month)

The effectiveness of the TIF will be assessed at the 8 study hospitals by measuring the use of key performance indicators during initial care of the injured before vs. after introduction of the TIF. Data on the key performance indicators will be obtained from observations by research assistants (RAs) of care provided by Emergency Health Service Providers (EHSPs) and by data from medical records. The investigators will obtain written consent from the EHSPs whose actions will be observed.

The investigators will then station RAs in the emergency units of recruited hospitals to observe EHSP practices regarding initial care of the injured using an observation form (derived from the TIF) as the investigators observe EHSPs assess and manage each participant arriving during the 8-hour shift of the RAs. The RAs will fill the form without interaction with EHSPs or the participant. For any components of the assessment and management that RAs are unable to directly observe, RAs will obtain information from the participants records to complete the observation form before the participant leaves the emergency unit.

After introduction of the TIF, RAs will complete the observation form for each participant as before. Prior to the participant leaving the emergency unit, RAs will make a blinded copy of the TIF completed by the EHSP in assessing and managing the participant. RAs will complete the observation form with information from participants records and/or from the EHSP-filled TIF. Both before and after introduction of the TIF, RAs will review the medical records of all participants observed for additional safety-related data, including occurrence of complications or death. These details will also be obtained from medical records at time of discharge for all participants who are admitted to the hospital.

The investigators will employ a stepped-wedge design in sequentially introducing the TIF to the 8 selected hospitals considered as 4 groups of 2 hospitals each. First, following 14 weeks of initial observation of EHSP practices at all 8 selected hospitals, the investigators will conduct a training workshop for EHSPs of the first randomly-selected group of hospitals on use of the TIF. Following the workshop, the EHSPs will be encouraged to begin use of the TIF at their hospitals. After another 14 weeks, the investigators will conduct the two-day training workshop for the next group of randomly selected hospitals, after which use of the TIF will begin at those hospitals. The investigators will continue this sequential conduct of training workshops followed by use of TIF every 14 weeks until all 8 hospitals have been exhausted. The RAs will continue to observe EHSP practices for a further 14 weeks during which the TIF will be in use at all 8 hospitals. The total duration of observation of EHSP practices will be 70 weeks. At the end of year one, the investigators will organize a one-day workshop for leadership of participating hospitals to review study progress.

ELIGIBILITY:
Inclusion Criteria:

* Emergency health care providers at the study hospitals
* Patient with injury who is treated in the emergency unit of one of the study hospitals

Exclusion Criteria:

* Non-emergency health care providers at the study hospitals
* Non-injured patient at the study hospitals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4105 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Donkor, Study Director — Kwame Nkrumah University of Science and Technology
Locations (1):
- Kwame Nkrumah University of Science and Technology, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gyedu A, Issaka A, Donkor P, Mock C. Utilization of a Trauma Quality Improvement Tool in a Clinical Trial: Effects When Tool Not Used. World J Surg. 2025 Jul;49(7):1960-1968. doi: 10.1002/wjs.12633. Epub 2025 May 19. PMID 40387168
- [Derived] Gyedu A, Amponsah-Manu F, Mensah S, Donkor P, Mock C. An evaluation of the Hawthorne effect in a clinical trial of trauma care in Ghana. World J Surg. 2024 Dec;48(12):3020-3026. doi: 10.1002/wjs.12410. Epub 2024 Nov 8. PMID 39516191
- [Derived] Gyedu A, Amponsah-Manu F, Awuku K, Ameyaw E, Korankye KK, Donkor P, Mock C. Differences in trauma care between district and regional hospitals and impact of a trauma intake form with decision support prompts in Ghana: A stepped-wedge cluster randomized trial. World J Surg. 2024 Mar;48(3):527-539. doi: 10.1002/wjs.12082. Epub 2024 Feb 5. PMID 38312029
- [Derived] Gyedu A, Stewart BT, Nakua E, Donkor P. Standardized trauma intake form with clinical decision support prompts improves care and reduces mortality for seriously injured patients in non-tertiary hospitals in Ghana: stepped-wedge cluster randomized trial. Br J Surg. 2023 Oct 10;110(11):1473-1481. doi: 10.1093/bjs/znad253. PMID 37612450

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process is complete. Recruitment was done at ERs of 8 participating hospitals from October 1, 2020 to March 31, 2022.
Pre-assignment Details: New participants were enrolled for every period within a sequence. The number of participants enrolled in each Period of the stepped wedge varied but add up to a total of 4,105.
  4,077 enrolled participants had complete primary data for analysis.
Units Other Than Participants: Hospitals
Groups:
- Sequence 1 (Hospitals 1&2): Hospitals were assigned to 14 weeks of initial observation (period 1), then 56 weeks of observation after introduction of the Trauma Intake Form (TIF) (periods 2-5).
  Patients were observed ONLY for their duration of stay in the hospital, NOT for the entire study duration.
- Sequence 2 (Hospitals 3&4): Hospitals were assigned to 28 weeks of initial observation (period 1 and 2), then 42 weeks of observation after introduction of the Trauma Intake Form (TIF) (periods 3-5).
  Patients were observed ONLY for their duration of stay in the hospital, NOT for the entire study duration.
- Sequence 3 (Hospitals 5&6): Hospitals were assigned to 42 weeks of initial observation (period 1-3), then 28 weeks of observation after introduction of the Trauma Intake Form (TIF) (periods 4 and 5).
  Patients were observed ONLY for their duration of stay in the hospital, NOT for the entire study duration.
- Sequence 4 (Hospitals 7&8): Hospitals were assigned to 56 weeks of initial observation (period 1-4), then 14 weeks of observation after introduction of the Trauma Intake Form (TIF) (periods 5).
  Patients were observed ONLY for their duration of stay in the hospital, NOT for the entire study duration.
Period: Period 1: 0-14 Weeks
Arm/Group | Sequence 1 (Hospitals 1&2) | Sequence 2 (Hospitals 3&4) | Sequence 3 (Hospitals 5&6) | Sequence 4 (Hospitals 7&8)
Started | 377; 2 Hospitals | 270; 2 Hospitals | 235; 2 Hospitals | 107; 2 Hospitals
Completed | 370; 2 Hospitals | 268; 2 Hospitals | 230; 2 Hospitals | 106; 2 Hospitals
Not Completed | 7; 0 Hospitals | 2; 0 Hospitals | 5; 0 Hospitals | 1; 0 Hospitals
Not completed — Incomplete Data | 7 | 2 | 5 | 1
Period: Period 2: 14-28 Weeks
Arm/Group | Sequence 1 (Hospitals 1&2) | Sequence 2 (Hospitals 3&4) | Sequence 3 (Hospitals 5&6) | Sequence 4 (Hospitals 7&8)
Started | 186; 2 Hospitals | 279; 2 Hospitals | 265; 2 Hospitals | 79; 2 Hospitals
Completed | 186; 2 Hospitals | 278; 2 Hospitals | 264; 2 Hospitals | 79; 2 Hospitals
Not Completed | 0; 0 Hospitals | 1; 0 Hospitals | 1; 0 Hospitals | 0; 0 Hospitals
Not completed — Incomplete Data | 0 | 1 | 1 | 0
Period: Period 3: 28-42 Weeks
Arm/Group | Sequence 1 (Hospitals 1&2) | Sequence 2 (Hospitals 3&4) | Sequence 3 (Hospitals 5&6) | Sequence 4 (Hospitals 7&8)
Started | 261; 2 Hospitals | 274; 2 Hospitals | 287; 2 Hospitals | 104; 2 Hospitals
Completed | 259; 2 Hospitals | 274; 2 Hospitals | 281; 2 Hospitals | 104; 2 Hospitals
Not Completed | 2; 0 Hospitals | 0; 0 Hospitals | 6; 0 Hospitals | 0; 0 Hospitals
Not completed — Incomplete Data | 2 | 0 | 6 | 0
Period: Period 4: 42-56 Weeks
Arm/Group | Sequence 1 (Hospitals 1&2) | Sequence 2 (Hospitals 3&4) | Sequence 3 (Hospitals 5&6) | Sequence 4 (Hospitals 7&8)
Started | 250; 2 Hospitals | 186; 2 Hospitals | 169; 2 Hospitals | 87; 2 Hospitals
Completed | 248; 2 Hospitals | 186; 2 Hospitals | 169; 2 Hospitals | 87; 2 Hospitals
Not Completed | 2; 0 Hospitals | 0; 0 Hospitals | 0; 0 Hospitals | 0; 0 Hospitals
Not completed — Incomplete Data | 2 | 0 | 0 | 0
Period: Period 5: 56-70 Weeks
Arm/Group | Sequence 1 (Hospitals 1&2) | Sequence 2 (Hospitals 3&4) | Sequence 3 (Hospitals 5&6) | Sequence 4 (Hospitals 7&8)
Started | 227; 2 Hospitals | 182; 2 Hospitals | 226; 2 Hospitals | 54; 2 Hospitals
Completed | 227; 2 Hospitals | 182; 2 Hospitals | 225; 2 Hospitals | 54; 2 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals | 1; 0 Hospitals | 0; 0 Hospitals
Not completed — Incomplete Data | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of 2,090 patients were enrolled before TIF introduction and 2,015 after TIF introduction, 23 patients and 5, respectively were excluded due to incomplete primary outcome data.
Groups:
- Pre TIF Introduction: Injured patients initially assessed and managed by emergency health service providers prior to introduction of the trauma intake form
- Post TIF Introduction: Injured patients initially assessed and managed by emergency health service providers after introduction of the trauma intake form
- Total: Total of all reporting groups
Arm/Group | Pre TIF Introduction | Post TIF Introduction | Total
Number analyzed (Participants) | 2067 | 2010 | 4077
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 453 | 419 | 872
  Between 18 and 65 years | 1407 | 1501 | 2908
  >=65 years | 207 | 90 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (16) | 30 (16) | 29 (16)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were 20 patients whose sex was not indicated before TIF and 4 patients whose sex was not indicated after TIF.
  Participants
    number analyzed (Participants) | 2047 | 2006 | 4053
    Female | 517 | 526 | 1043
    Male | 1,530 | 1,480 | 3010
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2067 | 2010 | 4077
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Appropriate Use of Key Performance Indicators in Initial Assessment and Management of the Injured at Non-tertiary Hospitals in Ghana
Description: The percentage of injured patients for whom key performance indicated eg. (Blood pressure, heart rate, oxygen saturation etc. ) are measured at initial assessment by emergency health service providers.
Time Frame: 17.5 months
Population: Spine immobilized was indicated only for RTI or fall victims Tetanus considered was only indicated for parties with for bites, burns, lacerations, aord abrasions
Measure: Count of Participants; unit: Participants
Arm/Group | Pre TIF Introduction | Post Introduction of TIF
Number analyzed (Participants) | 2067 | 2010
Participants
  Mobility at EU arrival assessed | 1807 | 1894
  Respiratory rate at EU arrival assessed | 1194 | 1787
  Airway assessed | 1506 | 1978
  Chest examined | 1284 | 1945
  Intra-abdominal bleeding evaluated | 747 | 1776
  Spine immobilized for RTI or fall victims: number analyzed (Participants) | 1453 | 1436
  Spine immobilized for RTI or fall victims | 250 | 1237
  Tetanus considered for bites, burns, lacerations, and abrasions: number analyzed (Participants) | 1654 | 1636
  Tetanus considered for bites, burns, lacerations, and abrasions | 1241 | 1434
  Date of injury recorded | 2012 | 1996
  Time of injury recorded | 1969 | 1454
  Important clinical data documented | 1083 | 1542
  Death | 47 | 22
Statistical Analysis 1: Comparison: Pre TIF Introduction vs Post Introduction of TIF; For mobility on EU arrival assessed,; Test type: Superiority — Power calculation - Expected enrollment: 25 patients/hospital/month, giving a total of 3,500 patients across all hospitals over 17.5 months. With an alpha of 0.05 and baseline TIF adherence rate of 50%, there was 80% power to detect 8.1-8.6% difference in KPI performance with 0.15-0.40 range in COV; p = 0.504, generalized linear mixed regression mode — Adjusted for TIF introduction and time periods as fixed effects and hospitals and time periods as random effects; Odds Ratio (OR) = 1.54
Statistical Analysis 2: Comparison: Pre TIF Introduction vs Post Introduction of TIF; Respiratory rate at EU assessed; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.169, generalized linear mixed regression mode; Odds Ratio (OR) = 2.31
Statistical Analysis 3: Comparison: Pre TIF Introduction vs Post Introduction of TIF; Airway assessed; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.006, generalized linear mixed regression; Odds Ratio (OR) = 25.29
Statistical Analysis 4: Comparison: Pre TIF Introduction vs Post Introduction of TIF; Chest examined; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.001, generalized linear mixed regression; Odds Ratio (OR) = 38.38
Statistical Analysis 5: Comparison: Pre TIF Introduction vs Post Introduction of TIF; For Intra-abdominal bleeding evaluated; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.001, generalized linear mixed regression; Odds Ratio (OR) = 93.01
Statistical Analysis 6: Comparison: Pre TIF Introduction vs Post Introduction of TIF; For Spine Immobilized for RTI or Fall Victims; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.001, generalized linear mixed regression; Odds Ratio (OR) = 354.91
Statistical Analysis 7: Comparison: Pre TIF Introduction vs Post Introduction of TIF; Splinting of Fractures Considered; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.001, generalized linear mixed regression; Odds Ratio (OR) = 4.95
Statistical Analysis 8: Comparison: Pre TIF Introduction vs Post Introduction of TIF; Tetanus Considered for bites, burns, lacerations, and abrasions; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.006, generalized linear mixed regression; Odds Ratio (OR) = 5.18
Statistical Analysis 9: Comparison: Pre TIF Introduction vs Post Introduction of TIF; Date of Injury Recorded; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.047, generalized linear mixed regression; Odds Ratio (OR) = 0.03
Statistical Analysis 10: Comparison: Pre TIF Introduction vs Post Introduction of TIF; Death; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.166, generalized linear mixed regression; Odds Ratio (OR) = 0.42
Statistical Analysis 11: Comparison: Pre TIF Introduction vs Post Introduction of TIF; Important Clinical Data Document; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.013, generalized linear mixed regression; Odds Ratio (OR) = 2.14

2. Secondary Outcome: Mortality
Description: All cause in-hospital mortality
Time Frame: Patients were followed for mortality until 18 months, when the last enrolled patient left hospital
Population: Injured patients initially assessed and managed at emergency units of select Ghanaian non-tertiary hospitals in Ghana
Measure: Count of Participants; unit: Participants
Groups:
- Mortality Pre-TIF Introduction: Patients who died at the study hospitals after presenting to the hospital in the period before TIF introduction. All 2,067 patients in this arm were at risk
- Mortality Post-TIF Introduction: Patients who died at the study hospitals after presenting to the hospital in the period after TIF introduction. All 2,010 patients in this arm were at risk
Arm/Group | Mortality Pre-TIF Introduction | Mortality Post-TIF Introduction
Number analyzed (Participants) | 2067 | 2010
Participants | 47 | 22
Statistical Analysis 1: Comparison: Mortality Pre-TIF Introduction vs Mortality Post-TIF Introduction; Test type: Superiority; p = 0.166, generalized linear mixed regression; Odds Ratio (OR) = 0.42

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events until 18 months, when the last enrolled patient left hospital
Description: By the nature of their conditions, all 4,077 enrolled injured patients were at risk of death and serious adverse events.
Groups:
- Mortality Pre-TIF Introduction: Patients who died at the study hospitals before TIF introduction. All 2,067 patients in this arm were at risk
- Mortality Post-TIF Introduction: Patients who died at the study hospitals after TIF introduction. All 2,010 patients in this arm were at risk
Arm/Group | Mortality Pre-TIF Introduction | Mortality Post-TIF Introduction
All-Cause Mortality (participants affected / at risk) | 47/2067 | 22/2010
Serious Adverse Events (participants affected / at risk) | 24/2067 | 6/2010
Other Adverse Events (participants affected / at risk) | 0/2067 | 0/2010
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mortality Pre-TIF Introduction (N=2067) | Mortality Post-TIF Introduction (N=2010)
wound infection (Infections and infestations) | 16 (16) | 6 (6) — wound infection as indicated by health providers in the medical records. The records were reviewed for complications at the time of discharge
pneumonia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0) — pneumonia as indicated by health providers in the medical records. The records were reviewed for complications at the time of discharge

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT04547192/Prot_SAP_000.pdf